CLINICAL TRIAL: NCT05131919
Title: Pembrolizumab for Locally Advanced, Irresectable, Non-metastatic dMMR Colorectal Cancers. The PUMA Study
Brief Title: Pembrolizumab for Locally Advanced, Irresectable, Non-metastatic dMMR Colorectal Cancers
Acronym: PUMA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N21PMA
Record Dates: First submitted 2021-11-02; First posted 2021-11-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single arm, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- pembrolizumab (Experimental): Treatment with pembrolizumab 200 mg.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Treatment with pembrolizumab 200 mg intravenously on day 1 of each 3-week cycle. Treatment will be continued for a maximum duration of 2 years, or until the tumor becomes resectable.
  Other Names: Keytruda

SUMMARY:
In this study, the efficacy of pembrolizumab in patients with locally advanced, irresectable dMMR colorectal cancer will be assessed.

DETAILED DESCRIPTION:
In this single-center, single arm, open-label, phase II study assessing the efficacy of pembrolizumab in patients with locally advanced, irresectable dMMR colorectal cancer, 25 patients will be enrolled. All patients will be treated with pembrolizumab 200 mg intravenously on day 1 of each 3-week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients at least 18 years of age
* Locally advanced, irresectable adenocarcinoma of the colon or rectum, not amenable to surgery, or for which induction therapy is required to reconsider surgery, or where free margins can only be obtained by major extension of the surgical procedure, as defined by one of the following:

  * Invasion of the duodenum, stomach, spleen or pancreatic head, for which major extension of the surgical procedure would be required to obtain free margins, and/or for which the chances of positive resection margins are high
  * Invasion or encasement of major blood vessels (superior mesenteric vessels, iliac vessels, portal vein)
  * Invasion or encasement of the ureter
* No signs of distant metastases on CT-scan and physical examination; patients may not be eligible for first-line treatment with pembrolizumab according to SoC
* Patients may not be eligible for standard of care first-line pembrolizumab for metastatic disease
* Patients may not be potentially eligible for the NICHE study: patients with primarily resectable disease, for which relatively minor extension of the procedure is required to achieve free margins, such as but not limited to a small bowel segment, abdominal wall
* ECOG performance status of 0 or 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention
* Screening laboratory tests must meet the criteria as defined in Table 1 and should be obtained within 10 days prior to the start of study intervention:

Absolute neutrophil count (ANC) ≥1500/µL; Platelets ≥100 000/µL; Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L, Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN; Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN; AST (SGOT) and ALT (SGPT) ≤2.5 × ULN; International normalized ratio (INR) OR prothrombin time (PT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants; Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

* A male participant must agree to use a contraception as detailed in Appendix 2 of this protocol during the treatment period and for at least 200 days (90 days plus the time required for pembrolizumab to undergo five half-lives) after the last dose of study treatment and refrain from donating sperm during this period.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to registration (see appendix 2). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* A female participant is eligible to participate if she is not pregnant (see appendix 2), not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) as defined in appendix 2 OR
  * A WOCBP who agrees to follow the contraceptive guidance in appendix 2 during the treatment period and for at least 120 days (30 days plus the time required for pembrolizumab to undergo five half lives) after the last dose of study treatment.
* CT-scan must be performed within 28 days prior to registration

Exclusion Criteria:

* Previous treatment with immune checkpoint inhibitors targeting including but not limited to CTLA-4, PD-1 or PD-L1
* Previous treatment with chemotherapy for the disease under study
* Prior radiotherapy for the disease under study
* Prior radiotherapy for other indications than the disease under study within 2 weeks of start of study intervention. Participants must have recovered from al radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* Intercurrent illnesses, including but not limited to infections, unstable angina pectoris
* Known history of Human Immunodeficiency Virus (HIV) infection and known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Underlying medical conditions that, in the investigator's opinion, will make the administration of the study drug hazardous or obscure the interpretation of toxicity determination of adverse events
* Active autoimmune disease requiring systemic treatment in the past 2 years;, or other medical conditions requiring systemic steroid or immunosuppressive medications, Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Diagnosis of immunodeficiency or conditions requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Live vaccines in the 4 weeks prior to inclusion
* History of uncontrolled medical or psychiatric illness
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Current pregnancy or breastfeeding
* Active malignancies other than disease under study within 3 years prior to inclusion, except for malignancies with a negligible recurrence rate (e.g. <10% in 5 years)
* Allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of pembrolizumab in patients with locally advanced, irresectable dMMR colorectal cancers by objective response rate (ORR) | 2.5 years
  ORR according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
To assess the major pathological response (MPR) in patients undergoing surgery | 2.5 years
  MPR is defined as < 10% residual viable tumor
To find biomarkers and evaluation strategies able to accurately assess complete and near-complete responses in order to pursue organ-sparing treatment | 2.5 years
  Association between changes in circulating tumor (ct)DNA and complete and near-complete responses, and risk of relapse
In case of surgery, to assess post-surgical outcome and infectious complications following neoadjuvant immunotherapy | 2.5 years
  Post-surgical outcome will be assessed by pathologic evaluation, infection complications will be graded according to CTCAE V5.0
To assess the date of relapse | 2.5 years
  As determined by disease recurrence or disease-related death during follow-up after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Chalabi, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No